CLINICAL TRIAL: NCT07310940
Title: THE EFFECT OF CHATBOT USE ON NURSING STUDENTS' CONCEPT MAP CONSTRUCTION SKILLS: A RANDOMIZED CONTROLLED STUDY
Brief Title: CHATBOT USE ON NURSING STUDENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Eda Ayten Kankaya, Asst. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9662
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-06

CONDITIONS: to Examine the Effect of Chatbot Use on Nursing Students
Keywords: Nurse education, Concept mapping, Nursing Students, Artificial Intelligence, Qualitative, Randomized controlled study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot-assisted concept mapping (Experimental): Students in this group received standard theoretical instruction on postoperative nursing care of cardiac surgery patients and, in addition, participated in a 15-minute training session on the use of ChatGPT and effective prompt techniques. During case-based learning activities, students were instructed to use the chatbot as a supportive tool while constructing concept maps.
  Interventions: Behavioral: Chatbot-assisted concept mapping
- Control group (Active Comparator): Students in this group received the same theoretical instruction on postoperative nursing care of cardiac surgery patients as the intervention group. They constructed case-based concept maps using textbooks, lecture notes, and course materials only, without the use of any chatbot or artificial intelligence-based tools.
  Interventions: Behavioral: Traditional concept mapping -Control Group

INTERVENTIONS:
Behavioral: Chatbot-assisted concept mapping — In this study, pre-test and post-test assessments were administered to students in both the intervention and control groups. Data were collected using the Student Information Form, Concept Map Evaluation Checklist, Attitude Toward Concept Mapping Scale, and a postoperative nursing care knowledge test.
  Students in the intervention group received training on ChatGPT use and prompt formulation and utilized the chatbot during the creation of case-based concept maps. The control group completed the same concept mapping activities using traditional learning resources without chatbot support.
  Arms: Chatbot-assisted concept mapping
Behavioral: Traditional concept mapping -Control Group — Students in the control group received the same theoretical instruction on postoperative nursing care of cardiac surgery patients. They constructed case-based concept maps using textbooks, lecture notes, and course materials only, without the use of any chatbot or artificial intelligence-based tools.
  Arms: Control group

SUMMARY:
Concept maps are visual tools that help students organize information and understand how ideas are related to each other. Although concept mapping is widely used in nursing education, many nursing students find it difficult to create effective concept maps. Recently, artificial intelligence tools such as ChatGPT have begun to be used in education and may help support students during learning activities. However, it is not yet clear whether using chatbots improves students' ability to create concept maps. This study aimed to examine whether using a chatbot (ChatGPT) helps nursing students develop better concept map construction skills. The study was conducted as a randomized controlled trial with second-year nursing students taking a surgical nursing course during the 2024-2025 spring semester. A total of 108 students were randomly assigned to either an intervention group or a control group. All students received the same theoretical education about postoperative care of cardiac surgery patients from the same instructor. Students in the intervention group received brief training on how to use ChatGPT and were allowed to use the chatbot while creating case-based concept maps. Students in the control group created concept maps using only textbooks and course materials. Students' knowledge, concept map quality, and attitudes toward concept mapping were evaluated. The results showed no significant difference between the two groups in terms of postoperative care knowledge or overall concept map scores. However, students who used ChatGPT had more positive attitudes toward concept mapping. Students also reported that the chatbot helped them understand complex information more easily and supported them during the concept map creation process.In conclusion, using a chatbot did not improve concept map performance scores, but it had a positive effect on students' attitudes and learning experiences. Chatbot-assisted learning may be a useful supportive tool in nursing education. Further studies with larger groups of students and longer follow-up periods are needed to better understand its effects on learning outcomes.

ELIGIBILITY:
Inclusion Criteria:

* -Taking the surgical nursing course for the first time

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Concept Map Construction Skill | Baseline (post-test), after the intervention - assessed once immediately after to the intervention.
  Concept Map Assessment Keys: Concept Map Assessment Keys are one of the tools used to evaluate concept maps. In this assessment tool, the student is evaluated on identifying a concept related to the topic and establishing meaningful connections between them, with 1 point awarded for each meaningful relationship/connection found. Another item evaluated is whether the student follows a hierarchical order according to priority when moving from general concepts/elements to more specific concepts, with 5 points awarded for each hierarchy established by the student. The student is awarded 10 points for each cross-connection established when moving from one concept section/group to another with a hierarchically meaningful connection.

SECONDARY OUTCOMES:
Attitude Toward the Concept Mapping Method | After the intervention - assessed once immediately after the intervention.
  Attitude Scale Towards the Concept Map: This will be used to assess the attitudes of all groups towards the concept map method prior to the initiative. It is a 5-point Likert-type scale developed to determine individuals' attitudes towards the concept map method. The scale consists of a total of 23 items and has a two-factor structure. The first factor consists of positive attitude items and contains 13 items. The second factor consists of negative attitude items and contains 10 items. Items on the scale are scored from 1 to 5. For positive items, the response "Strongly Agree" receives the highest score (5), while the response "Strongly Disagree" receives the lowest score (1). For negative items, the scoring is reversed; the response "Strongly Agree" receives the lowest score (1), while the response "Strongly Disagree" receives the highest score (5). As the total score obtained from the scale increases, the individual's attitude towards the concept mapping method is considered more po
Knowledge Level of Postoperative Nursing Care in Cardiac Surgery | Baseline (pre-test), before the intervention - assessed once immediately prior to the intervention.
  Cardiac Surgery Patient Nursing Care Knowledge Test: Prepared to measure student nurses' knowledge levels regarding post-cardiac surgery patient care. The test covers topics such as methods for maintaining the stability of patients after sternotomy, signs of cardiac tamponade, and the most commonly used graft types in coronary artery bypass grafting surgery. Additionally, postoperative care processes such as the importance of early mobilization, practices that support sternum healing, and the purpose of using compression stockings are also addressed in the test questions. Furthermore, the knowledge level regarding critical issues such as patient groups at risk of wound infection, appropriate mobilization planning, and nursing interventions to prevent pulmonary complications is assessed, and the aim is to increase nurses' awareness of these processes (Durmaz Edeer & Kankaya, 2025). Five experts were consulted for content validity for the knowledge test. Based on the evaluations obtaine
Students' Perceptions of Chatbot Use in Concept Mapping | Post intervention immediately
  Qualitative data were collected from students in the intervention group using two open-ended questions exploring their opinions on the role of chatbot use in the learning process and its contribution to concept map construction. Responses were analyzed using thematic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University,, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol